CLINICAL TRIAL: NCT04797312
Title: Comparison of an Opioid-Free Anesthesia Protocol Versus Standard Practices on Early and Late Post-operative Recovery
Acronym: SOFA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOFA
Record Dates: First submitted 2021-02-10; First posted 2021-03-15 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia; Anesthesia; Adverse Effect; Opioid Analgesic Adverse Reaction; Post-Op Complication
Keywords: Anesthesia; Quality of recovery; patient centered outcome
MeSH Terms: conditions — Postoperative Complications | interventions — Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Masking Description: The arm allocation is open for the anesthesia team and caregivers but the patient is blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia (OFA) protocol (Experimental)
  Interventions: Drug: Opioid Free Anaesthesia protocol
- standard practice protocol based on the use of opioids (sufentanil or remifentanil) (Sham Comparator)
  Interventions: Drug: standard practice protocol based on the use of opioids (sufentanil or remifentanil)

INTERVENTIONS:
Drug: Opioid Free Anaesthesia protocol — The OFA protocol begins with a systematic preoperative premedication with clonidine, continues with an adapted intraoperative management without opioid administration, but associating several molecules (clonidine, magnesium, lidocaine, ketamine) and ends with a continued administration of xylocaine up to 1 hour postoperatively in PACU. The use of an opioid in preoperative or intraoperative phases is considered as a deviation from the protocol.
  To these different molecules, the use of hypnotic molecules left to the choice of the practitioner and a curare will be systematically associated.
  Arms: Opioid free anesthesia (OFA) protocol
Drug: standard practice protocol based on the use of opioids (sufentanil or remifentanil) — Standard anesthetic practices can be summed up as the combination of a hypnotic, a morphinic (sufentanil or remifentanil) and a curare. The use of ketamine is allowed.
  Arms: standard practice protocol based on the use of opioids (sufentanil or remifentanil)

SUMMARY:
Opioid-Free Anesthesia (OFA) is an anesthesia protocol that does not use morphine, and is increasingly used routinely. Indeed, this protocol would theoretically allow a better post-operative analgesic control, a lower incidence of post-operative complications (e.g. post-operative nausea and vomiting). In the end, it would also allow a better overall post-operative recovery and a decrease in the incidence of chronic post-operative pain.

Nevertheless, the literature is poor on this issue and no randomized controlled study has evaluated the effect of the use of this type of anesthesia protocol on postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Surgery lasting more than 90 minutes with planned use of morphine analgesics during post-operative hospitalization (outside the PACU stay),
* ENT surgery, plastic and reconstructive surgery, digestive and visceral surgery, urological surgery and gynecological surgery,
* Surgery that does not involve any bone procedure,
* Written consent of the patient,
* French-speaking patient, able to understand and answer a questionnaire,
* Social security affiliation

Exclusion Criteria:

* Pregnant, breastfeeding or parturient woman,
* Person deprived of liberty by judicial or administrative decision,
* A person who is subject to a legal protection measure,
* Person unable to express consent,
* BMI < 18 and > 39 kg/m2,
* Drug contraindications, in particular hypersensitivity to the active substances of one of the study drugs (in particular lidocaine hydrochloride or amide- or clonidine-linked local anaesthetics) or to one of the excipients,
* Porphyria,
* Heart failure or unstable coronary artery disease,
* bradyarrhythmia due to sinus node disease or conduction clock, or Adam-Stock's syndrome, not fitted,
* Hepatocellular insufficiency with TP < or =50%,
* Chronic renal failure with glomerular filtration < 60 ml/min.
* Long-term treatment with Imipraminics, Neuroleptics, Baclofen, and all other molecules at risk of QT prolongation,
* Uncontrolled epilepsy,
* Chronic treatment with beta-blockers,
* Need for induction in fast sequence,
* Severe psychiatric or cognitive disorder that interferes with the evaluation through questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
FQoR-15 score at 24 hours | 24 hours after surgery
  Value of the French Quality of Recovery-15 score (minimum value of 0 and maximum value of 150, with a higher score for a better outcome).
  The QoR-15 questionnaires will be completed by the patient himself whenever possible, who could be helped by a nurse blinded to the assignment group, or by phone if the patient has returned home.

SECONDARY OUTCOMES:
FQoR-15 score at 48 and 72 hours | 48 and 72 hours after surgery
  Value of the French Quality of Recovery-15 score (minimum value of 0 and maximum value of 150, with a higher score for a better outcome).
  The QoR-15 questionnaires will be completed by the patient himself whenever possible, who could be helped by a nurse blinded to the assignment group, or by phone if the patient has returned home.
Pain on effort at 6, 12, 24, 48 and 72 hours | 6, 12, 24, 48 and 72 hours after surgery
  Pain evaluated via a 11-item analogue scale (from 0 to 10, with 10 for the worst pain) assessed by a blinded nurse.
Opioid consumption | 7 days
  Amount of opioid consumption in the 7 days, assessed by a blinded investigator.
Proportion of patient with at least one POMS complication at 24, 48 and 72 hours | 24, 48 and 72 hours
  POMS complication as described in the Post-operative Morbidity Survey, assessed by a blinded investigator.
Surgeon satisfaction at day 1 | day 1
  satisfaction concerning the protocole evaluated via a 11-item analogue scale (from 0 to 10, with 10 for the worst pain)
anesthesiologist satisfaction at day 1 | day 1
  satisfaction concerning the protocole evaluated via a 11-item analogue scale (from 0 to 10, with 10 for the worst pain)
Incidence of hemodynamic, rhythmic and allergic complications at day 1 | day 1
  Hemodynamic tolerance: the need to introduce catecholamines intraoperatively, or the need to stop one of the treatments in the protocol for hemodynamic reasons, Rhythmic tolerance: episode of extreme bradycardia < 35 bpm or tachycardia > 140 bpm for more than 30 seconds, The occurrence of a hypersensitivity reaction or other adverse events attributable to the anesthesia protocol.
  The complications are collected by the anesthesia team.
Proportion of patients with chronic pain at 3 months | 3 months
  Proportion of patients with chronic pain at 3 months detecting with brief pain inventory, assessed by a blinded investigator.
Quality of life measured from EQ VAS (EQ-5D-3L) | 3 months
  The Quality of life is evaluated via EQ VAS (derivating from the 5-level EQ-5D version (EQ-5D-3L), by a blinded assessor. The value from this scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine'. The scale is rated from 0 to 100.
Proportion of neuropathic pain at 3 months | 3 months
  The proportion of patients reporting neuropathic pain is defined by the DN4 questionnaire by a phone call with a blinded investigator. If the score is equal to or greater than 4/10, we define the presence of neuropathic pain.
Proportion of respect of the allocated anesthesia protocol | 24 hours after surgery
  Respect of the allocated protocol by the anesthesia team: OFA protocol will be considered complete if at least two of the following drugs are used between ketamine, lidocaine, clonidine and magnesium sulfate, and if no intraoperative opioids are used; the standard group will be considered complete if lidocaine, clonidine or magnesium sulfate are not used intra-operatively.
  This outcome is collected by one of the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Léger, MD, Principal Investigator — Angers University Hospital
Locations (1):
- University Hospital of Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leger M, Campfort M, Cayla C, Parot-Schinkel E, Lasocki S, Rineau E. Validation of an alternative French version of the Quality of Recovery-15 Score: the FQoR-15. Br J Anaesth. 2020 Oct;125(4):e345-e347. doi: 10.1016/j.bja.2020.05.052. Epub 2020 Jul 9. No abstract available. PMID 32654751
- [Background] Mauermann E, Ruppen W, Bandschapp O. Different protocols used today to achieve total opioid-free general anesthesia without locoregional blocks. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):533-545. doi: 10.1016/j.bpa.2017.11.003. Epub 2017 Nov 24. PMID 29739542
- [Derived] Leger M, Pessiot-Royer S, Perrault T, Parot-Schinkel E, Costerousse F, Rineau E, Lasocki S. The effect of opioid-free anesthesia protocol on the early quality of recovery after major surgery (SOFA trial): study protocol for a prospective, monocentric, randomized, single-blinded trial. Trials. 2021 Nov 27;22(1):855. doi: 10.1186/s13063-021-05829-x. PMID 34838109